CLINICAL TRIAL: NCT03892382
Title: A Pilot Study of Repetitive Transcranial Magnetic Stimulation for Improvement of Apathy in Amyotrophic Lateral Sclerosis
Brief Title: Repetitive Transcranial Magnetic Stimulation as Therapy for Apathy in Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants were not able to stay near our center for two weeks
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JagiellonianU62
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; rTMS; apathy; depression
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Lethargy; Depression

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to real or placebo (sham) stimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham stimulation will be provided by holding the stimulating coil perpendicularly to the scalp, which assures similar impression as during active stimulation but prevents significant magnetic field to reach the brain tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Active Comparator): 10 hertz (Hz) rTMS will be administered over the left dorsolateral prefrontal cortex. Therapy will include 10 daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 120% of the resting motor threshold intensity will be elicited.
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — High frequency rTMS to induce the long term potentiation in the left dorsolateral prefrontal cortex.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterized by progressive loss of central and peripheral motor neurons. ALS leads to death usually within 3 to 5 years from the onset of the symptoms. Available treatment can prolong the disease duration but cannot modify the disease course. Apathy is a frequent complication of ALS, affecting up to 30% of patients and affecting negatively the survival. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity with confirmed beneficial effect on apathy in several neurologic and psychiatric conditions. The purpose of this study is to compare the effectiveness of rTMS in improving the apathy in patients with ALS with placebo stimulation.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterized by progressive loss of central and peripheral motor neurons. ALS leads to death usually within 3 to 5 years from the onset of the symptoms. Available treatment can prolong the disease duration but cannot modify the disease course. Apathy is a frequent complication of ALS, which negatively influences quality of life (caga et al. 2018) and is an independent poor prognostic factor for survival (Caga et al. 2016). Similarly, the depression is also a frequent complication of ALS. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity with confirmed beneficial effect on apathy in several neurologic and psychiatric conditions like mild cognitive impairment (Padala et al. 2018), stroke (Sasaki et al. 2017), Alzheimer disease (Nguyen et al. 2017) and schizophrenia (Prikryl et al. 2013). The purpose of this study is to compare the effectiveness of rTMS in improving the apathy in patients with ALS with placebo stimulation and - as a secondary outcome - depression in patients with ALS.

Intervention will include ten daily sessions of rTMS. In each session 3000 magnetic pulses will be administered over the left dorsolateral prefrontal cortex. Stimulation intensity will equal 120% of the motor threshold value for the right first dorsal interosseus.

Assessment of apathy and of depression and daily functioning will be made before and after therapy, as well as two and four weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or probable ALS according to el Escorial criteria (Brooks et al. 2000)
* Moderate or severe depression defined as the score in Beck's Depression Inventory ≥20
* Mini-Mental State Examination score ≥26

Exclusion Criteria:

* Psychiatric symptoms, which may negatively influence patient's tolerance and adherence to therapy
* Respiratory insufficiency and other complications od advanced stages of ALS, which may compromise patient's ability to undergo the study procedure
* Contraindications for rTMS as listed by the Guidelines of the International Federation of Clinical Neurophysiology (Rossi et al. 2009) i.e. seizure in the past, epilepsy, presence of magnetic material in the reach of magnetic field, pregnancy, likelihood to get pregnant, intracranial electrodes, cardiac pacemaker or intracardiac lines, frequent syncopes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Apathy Evaluation Scale Clinical Version after rTMS, total score, range 18 to 72 with higher values representing a worse outcome | Baseline rTMS, directly (on the same 1 day) after finishing rTMS
  Change from baseline score in Apathy Evaluation Scale Clinical Version to the measurement taken directly after finishing rTMS.
Apathy Evaluation Scale Clinical Version first follow up, total score, range 18 to 72 with higher values representing a worse outcome | Baseline rTMS, two weeks after finishing rTMS
  Change from baseline score in Apathy Evaluation Scale Clinical Version to the measurement taken two weeks after finishing rTMS.
Apathy Evaluation Scale Clinical Version second follow up, total score, range 18 to 72 with higher values representing a worse outcome | Baseline rTMS, four weeks after finishing rTMS
  Change from baseline score in Apathy Evaluation Scale Clinical Version to the measurement taken four weeks after finishing rTMS

SECONDARY OUTCOMES:
Lateral Sclerosis Functional Rating Scale-Revised after rTMS, total score, range 0 to 40 with higher values representing a better outcome | Baseline rTMS, directly (on the same 1 day) after finishing rTMS
  Change from baseline score in Lateral Sclerosis Functional Rating Scale-Revised to the measurement taken directly after finishing rTMS.
Lateral Sclerosis Functional Rating Scale-Revised first follow up, total score, range 0 to 40 with higher values representing a better outcome | Baseline rTMS, two weeks after finishing rTMS
  Change from baseline score in the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised to the measurement taken two weeks after finishing rTMS.
Lateral Sclerosis Functional Rating Scale-Revised second follow up, total score, range 0 to 40 with higher values representing a better outcome | Baseline rTMS, four weeks after finishing rTMS
  Change from baseline score in Lateral Sclerosis Functional Rating Scale-Revised to the measurement taken directly after finishing rTMS
Beck's Depression Inventory ater rTMS, total score, range 0 to 63, with higher values representing a worse outcome | Baseline rTMS, directly (on the same 1 day) after finishing rTMS
  Change from baseline score in the Beck's Depression Inventory to the measurement taken directly after finishing rTMS.
Beck's Depression Inventory first follow up, total score, range 0 to 63, with higher values representing a worse outcome | Baseline rTMS, two weeks after finishing rTMS
  Change from baseline score in the Beck's Depression Inventory to the measurement taken two weeks after finishing rTMS.
Beck's Depression Inventory second follow up, total score, range 0 to 63, with higher values representing a worse outcome | Baseline rTMS, four weeks after finishing rTMS
  Change from baseline score in the Beck's Depression Inventory to the measurement taken four weeks after finishing rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Antczak, MD, Principal Investigator — Department of Neurology, Jagiellonian University Medical College
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
After completing the study, the details of neurophysiologic diagnostics including motor threshold, the age and gender as well as individual scores of Mini-Mental State Examination, AES-C, Beck's Depression Inventory and Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised will be made available to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study is published.
Access Criteria: On request send by e-mail: jantczak@cm-uj.krakow.pl

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Caga J, Hsieh S, Highton-Williamson E, Zoing MC, Ramsey E, Devenney E, Ahmed RM, Kiernan MC. Apathy and its impact on patient outcome in amyotrophic lateral sclerosis. J Neurol. 2018 Jan;265(1):187-193. doi: 10.1007/s00415-017-8688-4. Epub 2017 Nov 30. PMID 29189922
- [Background] Caga J, Turner MR, Hsieh S, Ahmed RM, Devenney E, Ramsey E, Zoing MC, Mioshi E, Kiernan MC. Apathy is associated with poor prognosis in amyotrophic lateral sclerosis. Eur J Neurol. 2016 May;23(5):891-7. doi: 10.1111/ene.12959. Epub 2016 Jan 29. PMID 26822417
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Nguyen JP, Suarez A, Kemoun G, Meignier M, Le Saout E, Damier P, Nizard J, Lefaucheur JP. Repetitive transcranial magnetic stimulation combined with cognitive training for the treatment of Alzheimer's disease. Neurophysiol Clin. 2017 Feb;47(1):47-53. doi: 10.1016/j.neucli.2017.01.001. Epub 2017 Feb 1. PMID 28161090
- [Background] Padala PR, Padala KP, Lensing SY, Jackson AN, Hunter CR, Parkes CM, Dennis RA, Bopp MM, Caceda R, Mennemeier MS, Roberson PK, Sullivan DH. Repetitive transcranial magnetic stimulation for apathy in mild cognitive impairment: A double-blind, randomized, sham-controlled, cross-over pilot study. Psychiatry Res. 2018 Mar;261:312-318. doi: 10.1016/j.psychres.2017.12.063. Epub 2018 Jan 5. PMID 29331848
- [Background] Prikryl R, Ustohal L, Prikrylova Kucerova H, Kasparek T, Venclikova S, Vrzalova M, Ceskova E. A detailed analysis of the effect of repetitive transcranial magnetic stimulation on negative symptoms of schizophrenia: a double-blind trial. Schizophr Res. 2013 Sep;149(1-3):167-73. doi: 10.1016/j.schres.2013.06.015. Epub 2013 Jun 25. PMID 23810122
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Sasaki N, Hara T, Yamada N, Niimi M, Kakuda W, Abo M. The Efficacy of High-Frequency Repetitive Transcranial Magnetic Stimulation for Improving Apathy in Chronic Stroke Patients. Eur Neurol. 2017;78(1-2):28-32. doi: 10.1159/000477440. Epub 2017 Jun 3. PMID 28578330